CLINICAL TRIAL: NCT00020605
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Phase IIB Study of Oral Naloxone for the Treatment of Opioid-Induced Constipation in Patients With Chronic, Non-malignant Pain or Malignant Pain
Brief Title: Naloxone in Treating Constipation in Patients Who Are Receiving Opioids for Chronic Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000068671; P30CA006516 (NIH); DFCI-NAL-0597; BWH-1999-P-002415/10; BWH-97-08658; ROXANE-NAL-0597
Record Dates: First submitted 2001-07-11; First posted 2004-04-05 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2001-10

CONDITIONS: Constipation, Impaction, and Bowel Obstruction; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; constipation, impaction, and bowel obstruction
MeSH Terms: conditions — Constipation; Intestinal Obstruction | interventions — Naloxone

INTERVENTIONS:
Drug: naloxone hydrochloride

SUMMARY:
RATIONALE: Naloxone may be effective in treating constipation that may be caused by opioid pain medications such as morphine.

PURPOSE: Phase III trial to determine the effectiveness of naloxone in relieving constiption in patients who are receiving opioids for chronic pain.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the long-term safety and efficacy of oral naloxone in treating opioid-induced constipation in patients with chronic malignant or non-malignant pain.

OUTLINE: This is a multicenter study. Patients receive oral naloxone twice daily. Each patient receives an escalating dose until the minimum effective dose or the maximum dose allowed is reached. The minimum effective dose is defined as the dose at which a patient has at least 4 bowel movements within 7 days. Patients receive the minimum effective dose for 7 days and then continue long-term treatment for a maximum of 72 weeks. Patients receiving the maximum dose allowed with fewer than 4 bowel movements per week will discontinue study therapy.

PROJECTED ACCRUAL: Approximately 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Moderate to severe opioid-induced constipation Previously enrolled on protocols NAL-0396, NAL-0397, and/or NAL-0398 OR Low frequency of bowel movements, defined as fewer than 3 per week during the past 2 weeks, AND either of the following: Score of "some", "quite a bit", or "very much" on the constipation distress scale Laxative or enema dependence Daily opioid intake equivalent to at least 30 mg of oral morphine for chronic pain of malignant or non-malignant origin Stable dose of opioid analgesic agent for at least 2 weeks No score of "excruciating" on verbal pain scale No history of partial or complete bowel obstruction No constipation secondary to factors other than opioids (e.g., autonomic neuropathy or intra-abdominal adhesions)

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Potassium normal Other: No uncontrolled endocrinopathy or diabetes No psychiatric disorder or encephalopathy that would preclude study No clinically significant medical conditions that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Concurrent chemotherapy allowed provided patient has completed at least 1 course prior to study Endocrine therapy: Concurrent hormonal therapy allowed provided dosage is stable for at least 2 weeks prior to study Radiotherapy: No concurrent palliative radiotherapy to spine, abdomen, or pelvic area Surgery: Not specified Other: At least 30 days since other investigational drug

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Katz, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States